CLINICAL TRIAL: NCT03634722
Title: Beijing Key Laboratory of Female Pelvic Floor Disorders of Peking University People's Hospital
Brief Title: The Efficacy of Transcutaneous Electrical Nerve Stimulation on LUTS: One Prospective Study.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PKUPH2
Record Dates: First submitted 2018-07-23; First posted 2018-08-16 (Actual); Last update posted 2018-12-27 (Actual); Status verified 2018-12

CONDITIONS: Pelvic Organ Prolapse
Keywords: transcutaneous electrical nerve stimulation;
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: the transcutaneous electrical nerve stimulation by PHENIX4-8-8 PLUS
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The intervention group (Experimental): the transcutaneous electrical nerve stimulation by PHENIX4-8-8 PLUS
  Interventions: Device: PHENIX4-8-8 PLUS
- The observational group (No Intervention): routine nursing

INTERVENTIONS:
Device: PHENIX4-8-8 PLUS — transcutaneous electrical nerve stimulation by PHENIX4-8-8 PLUS
  Arms: The intervention group

SUMMARY:
The study is a prospective study at a single institution. Investigators create strict inclusion and exclusion criteria, selecting 126 patients who undergo the pelvic reconstructive surgery. 63 patients in the intervention group accept 10 times of the transcutaneous electrical nerve stimulation.

DETAILED DESCRIPTION:
All the patients have severe pelvic organ prolapse and undergo the pelvic reconstructive surgery. Investigators evaluate all patients' lower urinary tract symptoms, quality of life score, overactive bladder questionnaire, maximal rate and residual urine volume, at 1, 3, 6 and 12 months after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* severe pelvic organ prolapse(POP-Q:3/4 stage)
* accept pelvic reconstructive surgery

Exclusion Criteria:

* Dominant stress urinary incontinence
* Serious medical problems
* mental disease
* infectious disease

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2019-01-01 (Estimated); Primary Completion 2019-01-07 (Estimated); Study Completion 2020-12-11 (Estimated)

PRIMARY OUTCOMES:
the rate of urinary retention | three days after surgery
  urinary residual volume

SECONDARY OUTCOMES:
the rate of urinary incontinence | three days; seven days; one month; three months; six months after surgery
  according to the 1-h pad test

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Sun, Study Chair — Beijing Key Laboratory of Female Pelvic Floor Disorders
Locations (1):
- The Peking University People's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
The Transcutaneous Electrical Nerve Stimulation can decrease the rate of Lower Urinary Tract Symptoms after Pelvic Reconstructive Surgery
Supporting Information: Study Protocol, CSR
Time Frame: two years